CLINICAL TRIAL: NCT04392310
Title: Outcomes of Acute Myeloid Leukemia Patients in Assiut University Hospital
Brief Title: Outcomes of Acute Myeloid Leukemia Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Abdelsalam Abodeif sayed, Sohage_Tema, Assiut University
Other Study IDs: Outcomes of AML
Record Dates: First submitted 2019-09-27; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To assess overall survival of AML patient.
2. To measure rate of disease free survival.
3. rate of non relapse mortality.
4. rate of complete remission .
5. percentage of refractory disease.
6. percentage of relapsed disease.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a malignant disorder of the bone marrow which is characterized by malignant clonal expansion and differentiation arrest of myeloid progenitor cells.

The etiology of AML is heterogeneous. In some patients, prior exposure to therapeutic, occupational or environmental DNA-damaging agents is implicated, but most cases of AML remain without a clear etiology.

The incidence of AML had been higher than that of the other three subtypes of leukemia ( [ALL], [CML], and [CLL])& accounts for the highest percentage (62%) of leukemic deaths.

AML is primarily a disease of older adults. The age-adjusted incidence for those aged 65 years or older is 20.1 per 100,000 persones in comparison to 2.0 per 100,000 person-years for those younger than 65 years old.

Males are 1.2-1.6 times more likely to develop AML during their lifetime as evidenced by population-based studies in the US, UK, Canada, Denmark, Australia and Algeria. AML is one of the most common form of Hematological Malignancy in adults and has the shortest survival (5-year survival = 24%). Curative therapies, including intensive chemotherapy and allogeneic stem cell transplantation, are generally applicable to a minority of patients who are younger and fit, while most older individuals exhibit poor prognosis and survival. Differences in patient outcomes are influenced by disease characteristics, access to care including active therapies and supportive care, and other factors. After many years without therapeutic advances, several new therapies have been approved and are expected to impact patient outcomes, especially for older patients and those with refractory disease.

ELIGIBILITY:
Inclusion Criteria:

* AML patients, aged more than 18yrs and received chemotherapy (aggressive or palliative).

Exclusion Criteria:

* patients less than 18years old.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute myeloid leukemia patients outcomes
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the overall survival of AML patients. | One year
  Assessment of the overall survival of AML patients.

REFERENCES:
- [Background] De Kouchkovsky I, Abdul-Hay M. 'Acute myeloid leukemia: a comprehensive review and 2016 update'. Blood Cancer J. 2016 Jul 1;6(7):e441. doi: 10.1038/bcj.2016.50. PMID 27367478